CLINICAL TRIAL: NCT03460483
Title: Ohio Prevention and Treatment of Endometrial Cancer (OPTEC) Initiative: Universal Screening for DNA Mismatch Repair Deficiency and Personalized Cancer Treatment
Brief Title: Universal Endometrial Cancer DNA Sequencing for Detection of Lynch Syndrome and Personalized Care
Acronym: OPTEC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Paul Goodfellow, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: OSU-17149; NCI-2018-00218 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2018-03-01; First posted 2018-03-09 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Endometrial Adenocarcinoma; Endometrial Carcinoma; Lynch Syndrome; Relatives
MeSH Terms: conditions — Endometrial Neoplasms; Colorectal Neoplasms, Hereditary Nonpolyposis | interventions — Genetic Counseling; Genetic Testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Comprehensive LS genetic testing (Experimental): Testing for inherited forms of cancer and tumor sequencing
  Interventions: Other: Genetic Counseling; Other: Genetic Testing; Other: Laboratory Biomarker Analysis; Procedure: Mutation Carrier Screening

INTERVENTIONS:
Other: Genetic Counseling — Undergo genetic counseling
Other: Genetic Testing — Undergo genetic testing
  Other Names: genetic analysis; Genetic Examination; Genetic Test
Other: Laboratory Biomarker Analysis — Correlative studies
Procedure: Mutation Carrier Screening — Undergo tumor screening via next-generation sequencing

SUMMARY:
This clinical trial studies universal screening for deoxyribonucleic acid (DNA) mismatch repair deficiency in patients with endometrial cancer, mutations in the genes responsible for Lynch syndrome (inherited forms of endometrial cancers) and other DNA changes that could help guide treatment strategies. Universal tumor DNA sequencing may help doctors better understand how to personalize care, increase length of life, and increase quality of life in patients with endometrial cancer and their relatives.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Molecular classification of tumor abnormalities through innovative upfront next-generation DNA sequencing.

II. Identify endometrial cancer (EC) patients with inherited EC, specifically Lynch syndrome (LS), using both tumor and normal (blood) DNA testing.

III. Develop a comprehensive approach to genetic risk assessment and management including improved cascade testing in at-risk relatives.

IV. Provide local access to genetic counseling for patients with harmful germline mutations.

V. Identify molecular signatures that may be associated with favorable response to specific treatments (including chemotherapeutic agents, non-surgical options, and novel clinical trials [in particular, patients with mismatch repair (MMR)-deficient or POLE-mutant tumors]).

VI. Determine if recurrence likelihood can be predicted from molecular signature.

VII. Identify EC patients with select molecular signatures for recruitment to long-term follow-up, cancer prevention, and treatment studies.

OUTLINE:

Patients with endometrial cancer undergo clinical testing for inherited cancer mutations using blood DNA and via next-generation sequencing of tumor samples. Patients testing positive for Lynch syndrome or other cancer susceptibilities will undergo genetic counseling and testing and counseling will be offered to their family members.

ELIGIBILITY:
Inclusion Criteria:

* Adult women who had a hysterectomy or diagnostic biopsy proving endometrial adenocarcinoma (any stage) between 10/1/2017 and 4/30/2020, and received care at one of the participating hospitals
* Adult relatives of the EC patients found to have LS

Exclusion Criteria:

* Individuals must be able to speak and read English; non-English speaking individuals will be excluded
* Individuals must be able to consent for themselves; those who are unable to consent for themselves for any reason will be excluded
* Prisoners will be specifically excluded from participation in the study
* Women who have uterine sarcomas are excluded
* Pregnant women are not eligible for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1001 (Actual)
Dates: Start 2018-03-30 (Actual); Primary Completion 2025-06-15 (Actual); Study Completion 2025-06-15 (Actual)

PRIMARY OUTCOMES:
Incidence of endometrial cancer patients with Lynch syndrome | Up to 3 years
  Measured by molecular profiling of tumor deoxyribonucleic acid (DNA) via next-generation sequencing.
Incidence of tumors with microsatellite instability and/or somatic POLE mutations | Up to 3 years
  Measured by molecular profiling of tumor DNA via next-generation sequencing.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Goodfellow, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (9):
- United States (9):
  - Summa Akron City Hospital/Cooper Cancer Center, Akron, Ohio
  - Aultman Health Foundation, Canton, Ohio
  - University of Cincinnati, Cincinnati, Ohio
  - TriHealth Cancer Institute-Westside, Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Ohio Health, Columbus, Ohio
  - Mercy Health - St. Vincent Medical Center, Toledo, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu